CLINICAL TRIAL: NCT01668225
Title: Impact of Follicular and Blood G-CSF on Pregnangcy and Implantation Rate During Modified Natural in Vitro Fertility Cycle
Brief Title: Impact of Follicular and Blood G-CSF During a Natural Cycle of IVF
Acronym: GCSFnat
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: OVO-11-02
Record Dates: First submitted 2012-06-19; First posted 2012-08-20 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample Follicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- G-CSF FIV nat: Patient following a natural In Vitro Fecondation cycle
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Taking blood sample of the patient during the day 3, triggering day, oocyte collection day and pregnancy test day.
  Taking the follicular fluid during the oocyte collection day

SUMMARY:
Recently, scientists look into G-CSF (Granulocyte - Colony Stimulatin Factor). The use of this molecule is increasing in reproduction pathology. High level of follicular and blood G-CSF on the day of oocyte retrieval could correlate with higher pregnancy and implantation rates.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 43 years old
* Women natural In Vitro Fecondation

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a natural cycle of an In Vitro Fecondation
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Serum and / or follicular minimum level of G-CSF predictive of pregnancy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Ovo Fertilité, Montreal, Quebec, Canada